CLINICAL TRIAL: NCT03813797
Title: LaPAroscopic Low pRessure cOlorectal Surgery
Acronym: PAROS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHUBX 2018/42
Record Dates: First submitted 2019-01-08; First posted 2019-01-23 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Malignant or Benign Pathology
Keywords: Low Pressure; Laparoscopy; Colectomy; Pneumoperitoneum; AirSeal
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The study will be carried out:
  * Blind patient: The patient will not know the group he belongs to, in order to minimize the bias related to the self-evaluation of postoperative pain
  * Blind for the outpatient evaluator: the surgeon will blindly evaluate the primary endpoint: patient's discharge criteria. This "evaluator" surgeon will be different from the "operator" surgeon The blind will minimize the measurement bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Low Pressure (5-7 mmHg) (Experimental): Laparoscopic colectomy surgery with low pressure (5-7mmHg)
  Interventions: Device: Airseal®
- Arm B: Standard pressure (12-15 mmHg) (Active Comparator): Laparoscopic colectomy surgery with standard pressure (12-15mmHg)
  Interventions: Device: Standard Insufflation

INTERVENTIONS:
Device: Airseal® — Medical device set to the mode Airseal®, pressure adjustment between 5 and 7 mmHg
  Arms: Arm A: Low Pressure (5-7 mmHg)
Device: Standard Insufflation — Medical device set to the mode "Standard Insufflation", pressure adjustment between 12 and 15 mmHg
  Arms: Arm B: Standard pressure (12-15 mmHg)

SUMMARY:
Laparoscopy by its mini-invasive character has revolutionized abdominal and colorectal surgery but certain limitations remains (post-operative pain due to pneumoperitoneum, pneumoperitoneum stability, visibility during bleeding, smoke evacuation). The medical device for continuous pressure insufflation during laparoscopic procedures Airseal® would allow the maintenance of pneumoperitoneum at a lower pressure. The stable low pressure (7mmHg) is described in the literature for 15 years as the best way to reduce scapular pain, but until the marketing of Airseal, working at 7mmHg was not possible because the space of work was not stable. Moreover, this device makes it possible to obtain a better vision because of the evacuation of the fumes potentially leading to a reduction in the operating time.

DETAILED DESCRIPTION:
This research focuses on a medical device that allows the surgeon to perform the surgical procedure at a lower pressure than usual.

The main objective of this study is to compare the duration of hospitalization of patients with laparoscopic colectomy at low pressure (5-7 mmHg) versus standard pressure (12-15 mmHg) It is a prospective randomized monocentric double blind study

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Colonic resection (right or left) performed for benign or malignant pathology
* Laparoscopic procedure
* Informed consent signed
* Social Insurance

Exclusion Criteria:

* Laparotomy procedure
* Associated resection (except appendectomy or liver biopsy
* Emergency procedure
* Pelvic sepsis
* Pregnant or breast-feeding woman.
* Persons deprived of liberty or under guardianship
* Impossibility for compliance to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-05-25 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Length of postoperative hospital stay | From surgery to the end of the hospitalization (max 30 days)
  To determine the length of hospitalization

SECONDARY OUTCOMES:
Surgery time | During surgery
  To determine the surgery time
Appreciation of visual quality by surgeon | During surgery
  To determine the rate of visual quality during surgery: poor, medium or good quality
Impact of the use of microlaparoscopic instruments | During surgery
  To determine the rate of use of the microsurgery microlaparoscopic instruments (3mm)
Rates of conversion | During surgery
  Conversion to laparoscopy with standard pressure or conversion to laparotomy
Blood pressure (mmHg) | During surgery
  To examine the variation of blood pressure during surgery (at the beginning, middle and at the end)
Cardiac frequency (/ min) | During surgery
  To examine the variation of cardiac frequency during surgery (at the beginning, middle and at the end)
Volume replacement (mL) | During surgery
  To examine the volume replacement during surgery (at the beginning, middle and at the end)
Driving pressure (mmHg) | During surgery
  To examine the variation of drinving pressure during surgery (at the beginning, middle and at the end)
Oxygen saturation (%) | During surgery
  To examine the variation of SA02 (%) during surgery (at the beginning, middle and at the end)
Partial pressure of mean expired of carbon dioxide (mmHg) | During surgery
  To examine the variation PECO2 (mmHg) during surgery (at the beginning, middle and at the end)
Surgical and medical morbidity | From surgery until 30 days (max 45 days)
  To analyse the cumulative Clavien-Dindo at 30 days
Postoperative pain | 2 hours, 4 hours, 8 hours and 24 hours after the surgery
  Pain was evaluated with the Numeric Rating Scale (NRS, from 0 (no pain) to 10 (hurts worst)
Use of analgesics | An average of 5 days after the surgery
  To evaluate the rate of analgesics administrated (from step1 to step3)
Time before the passage of first stool (days) | An average of 5 days after the surgery
  To determine the delay of the laxation and gas response
Time before the passage of first gas (days) | An average of 5 days after the surgery
  To determine the delay of the gas response
Time before mobilization (Days before 1st time sitting and standing) | An average of 5 days after the surgery
  To determine the delay before mobilization
Quality of cancer surgery | During surgery
  Rate of curative surgery (R0)
Number of lymph nodes examed | During surgery
  Number of lymph nodes examed during a cancer surgery

CONTACTS AND LOCATIONS:
Overall Officials: Quentin DENOST, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Chu de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Celarier S, Monziols S, Celerier B, Assenat V, Carles P, Napolitano G, Laclau-Lacrouts M, Rullier E, Ouattara A, Denost Q. Low-pressure versus standard pressure laparoscopic colorectal surgery (PAROS trial): a phase III randomized controlled trial. Br J Surg. 2021 Aug 19;108(8):998-1005. doi: 10.1093/bjs/znab069. PMID 33755088